CLINICAL TRIAL: NCT06435806
Title: Advancing Medical Illustration in Patient Education Materials: From Art to Science. Study 1: Medical Illustration Design Characteristic Evaluation
Brief Title: Medical Illustration Design Characteristic Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Tufts Medical Center (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 427440
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: We will select 10 binary distinctions of medical illustration design elements and test each in a two-arm between-subjects evaluation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (20):
- Medical Illustration Design Distinction 1, version A (Experimental): Medical Illustration Design Distinction 1, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 1, version B (Experimental): Medical Illustration Design Distinction 1, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 2, version A (Experimental): Medical Illustration Design Distinction 2, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 2, version B (Experimental): Medical Illustration Design Distinction 2, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 3, version A (Experimental): Medical Illustration Design Distinction 3, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 3, version B (Experimental): Medical Illustration Design Distinction 3, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 4, version A (Experimental): Medical Illustration Design Distinction 4, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 4, version B (Experimental): Medical Illustration Design Distinction 4, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 5, version A (Experimental): Medical Illustration Design Distinction 5, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 5, version B (Experimental): Medical Illustration Design Distinction 5, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 6, version A (Experimental): Medical Illustration Design Distinction 6, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 6, version B (Experimental): Medical Illustration Design Distinction 6, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 7, version A (Experimental): Medical Illustration Design Distinction 7, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 7, version B (Experimental): Medical Illustration Design Distinction 7, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 8, version A (Experimental): Medical Illustration Design Distinction 8, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 8, version B (Experimental): Medical Illustration Design Distinction 8, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 9, version A (Experimental): Medical Illustration Design Distinction 9, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 9, version B (Experimental): Medical Illustration Design Distinction 9, version B
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 10, version A (Experimental): Medical Illustration Design Distinction 10, version A
  Interventions: Other: Medical Illustration design
- Medical Illustration Design Distinction 10, version B (Experimental): Medical Illustration Design Distinction 10, version B
  Interventions: Other: Medical Illustration design

INTERVENTIONS:
Other: Medical Illustration design — We will test 10 binary design variants for medical illustrations (for example, with and without cut-away, with and without text labels, etc). Specific variants to be identified during first task of project.

SUMMARY:
The goal of this study is to understand what people understand from medical illustrations, and what meaning and emotions (such as anxiety) they derive from different design elements.

DETAILED DESCRIPTION:
The investigators will conduct cognitive interviews to understand the meaning laypersons obtain from different illustrations, their opinions on illustration styles, and their level of anxiety after viewing illustrations.

The investigators will also study the effect of systematically varying medical illustration designs on layperson understanding and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Speaks English or Spanish ﬂuently
* Is able to independently consent
* Has adequate corrected vision to read patient education documents

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8200 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge | Baseline and 30 minutes
  A multiple-item knowledge test designed to test comprehension of the patient education document
State Anxiety scale from State-Trait Anxiety Inventory | 30 minutes
  Self-report state anxiety scale from the State-Trait Anxiety Inventory. 20 items, 4-point Likert scale. A higher score indicates more severe anxiety with a potential range from 20 to 80.

SECONDARY OUTCOMES:
Satisfaction with the medical illustration | 30 minutes
  Likert items to assess satisfaction with the document and illustration
Reading Effort | 30 minutes
  Likert items to assess perceived effort in reading a document and illustration
Acceptability | 30 minutes
  Likert items to assess acceptability and appropriateness of the illustration

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bickmore, PhD, Principal Investigator — Northeastern University
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Northeastern University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Transcripts from 100 cognitive interviews, and quantitative measures of comprehension and anxiety from 7,600 participant reactions to patient education documents will be generated. We will create de-identified data sets of all quantitative human subjects data that will be preserved and shared. The purpose for creating this is to allow other investigators access to the data to both validate our findings and to further advance inquiry in the field.
Supporting Information: Study Protocol, ICF
Time Frame: Prior to end of the study.
Access Criteria: Sharing of de-identified human subjects data will be consistent with HIPAA guidelines and the Final NIH Statement on Sharing Research Data. We do not anticipate any limitations on sharing.